CLINICAL TRIAL: NCT05395403
Title: Use of Automated Office Blood Pressure Monitoring in Older Working-age Adults
Brief Title: Use of Automated Office Blood Pressure Monitoring
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Collaborators: Troy University (Unknown)
Responsible Party: Principal Investigator, Tonya Breaux-Shropshire, Clinical Scientist and Transplant Cood, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: IRB-300006396
Record Dates: First submitted 2022-04-19; First posted 2022-05-27 (Actual); Last update posted 2022-05-27 (Actual); Status verified 2022-05

CONDITIONS: Hypertension; Uncontrolled Hypertension; Hypertension, White Coat; Hypertension, Resistant to Conventional Therapy
MeSH Terms: conditions — Hypertension; White Coat Hypertension; Hypertension Resistant to Conventional Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Office Blood Pressure Measurement (OBPM) (Experimental): Traditional office blood pressure monitoring in the primary care clinical environment.
  Interventions: Device: Blood pressure measurement device
- Automated Office Blood Pressure Measurement (AOBPM) (Experimental): Blood pressure measurement using a validated BpTRU device
  Interventions: Device: Blood pressure measurement device
- Home Blood Pressure Measurement (HBPM) (Experimental): Blood pressure measurement at patient's home using home monitoring device.
  Interventions: Device: Blood pressure measurement device

INTERVENTIONS:
Device: Blood pressure measurement device — The use of three different devices: traditional office blood pressure measurement cuff (OBPM), automated office blood pressure measurement cuff (AOBPM), and home blood pressure measurement cuff (HBPM).

SUMMARY:
Blood pressure measurements by three methods Office Blood Pressure Measurement (OBPM), Automated Office Blood Pressure Measurement (AOBPM), and Home Blood Pressure Measurement (HBPM) were collected retrospectively across three visits for patients (N=28) referred to a specialty hypertension (HTN) clinic. Demographic data were analyzed using summary statistics. The differences between AOBPM, HBPM, and OBPM were examined using mixed models repeated measures analysis for time and method for each visit.

ELIGIBILITY:
Inclusion Criteria:

* 19 years and older
* Uncontrolled BP
* Prescribed three or more antihypertensive medications at the time of referral
* Higher risk for poor CV outcomes than patients with essential HTN
* OBPM systolic BP of greater than 140 mmHg and diastolic BP of greater than or equal to 90 mm Hg upon initial clinic assessment.

Exclusion Criteria:

* Less than 19 years old
* Had a systolic BP of less than 140 mm Hg and diastolic BP of less than 90 mmHg upon initial clinic assessment.
* Also, patients on less than three antihypertensive medications, with less than three visits, and who have controlled OBPM were excluded.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2021-03-05 (Actual); Primary Completion 2021-07-05 (Actual); Study Completion 2021-07-05 (Actual)

PRIMARY OUTCOMES:
Number of participants using Traditional office blood pressure measurement (OBPM) | Baseline
  Blood pressure control: Traditional office blood pressure measurement less than 140/90 mm Hg
Number of participants using Traditional office blood pressure measurement (OBPM) | Up to 8 weeks
  Blood pressure control: Traditional office blood pressure measurement less than 140/90 mm Hg
Number of participants using Traditional office blood pressure measurement (OBPM) | Up to 16 weeks
  Blood pressure control: Traditional office blood pressure measurement less than 140/90 mm Hg
Number of participants using Automated office blood pressure measurement (AOBPM) | Baseline
  Blood pressure control: Automated office blood pressure measurement less than 130/80 mm Hg
Number of participants using Automated office blood pressure measurement (AOBPM) | Up to 8 weeks
  Blood pressure control: Automated office blood pressure measurement less than 130/80 mm Hg
Number of participants using Automated office blood pressure measurement (AOBPM) | Up to 16 weeks
  Blood pressure control: Automated office blood pressure measurement less than 130/80 mm Hg
Number of participants using Home blood pressure measurement (HBPM) | Baseline
  Blood pressure control: Home blood pressure measurement less than 130/80 mm Hg
Number of participants using Home blood pressure measurement (HBPM) | Up to 8 weeks
  Blood pressure control: Home blood pressure measurement less than 130/80 mm Hg
Number of participants using Home blood pressure measurement (HBPM) | Up to 16 weeks
  Blood pressure control: Home blood pressure measurement less than 130/80 mm Hg

CONTACTS AND LOCATIONS:
Locations (1):
- University of Alabama at Birmingham, Birmingham, Alabama, United States